CLINICAL TRIAL: NCT00645281
Title: Symptom Specific Effectiveness of Tolterodine ER 4 mg in Patients With Symptoms of Overactive Bladder (OAB) in a Primary Care Setting. A Phase IV, Open-label, Single-arm, Non-randomized, Trial in Adult Patients With OAB.
Brief Title: A Study to Evaluate the Efficacy of Tolterodine on Specific Symptoms in Adult Patients With Overactive Bladder.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6121001
Record Dates: First submitted 2008-03-25; First posted 2008-03-27 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive

ARMS (1):
- tolterodine ER group (Experimental)
  Interventions: Drug: tolterodine extended release

INTERVENTIONS:
Drug: tolterodine extended release — Tolterodine ER capsule 4 mg daily for 12 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tolterodine in impacting the primary symptom or complaint of patients with OAB.

ELIGIBILITY:
Inclusion Criteria:

* self-reported symptoms of OAB for ≥ 3 months prior to screening
* OAB as defined by urinary frequency (a minimum of 8 micturitions per 24 hours)
* urgency (defined as a strong and sudden desire to urinate) or urge incontinence a minimum of 2 episodes in 3 days, as confirmed by the micturition diary between screening and baseline
* patients who describe the degree of bothersomeness of their most bothersome OAB symptom as "moderately ", "a great deal ", or "a very great deal" per the OAB Bother Rating Scale

Exclusion Criteria:

* any condition that would contraindicate their usage of tolterodine once daily, including: narrow angle glaucoma, urinary retention, gastric retention
* any clinically significant local urinary tract pathology which could mimic the symptoms of OAB, such as infection or hematuria
* stress incontinence, functional, or overflow incontinence as determined by the investigator
* symptomatic acute urinary tract infection (UTI) during the run-in period, or recurrent UTIs defined by treatment for symptomatic UTI >3 times in the 12 months prior to participation in this clinical trial
* clinically significant urinary tract obstruction
* history of lower urinary tract surgery (e.g. prostate removal or destruction, incontinence surgery) within the past 3 months
* clinically significant interstitial cystitis or significant bladder pain syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 896 (Actual)
Dates: Start 2004-03; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 12 in the micturition bladder diary variable related to the primary symptom of the patient at the time of study entry | 12 weeks

SECONDARY OUTCOMES:
OAB Bother Rating Scale at baseline | baseline
Change from baseline to Week 4 and 12 in micturition bladder diary variables | 12 weeks
Change from baseline to Week 4 and 12 in Patient's Perception of Bladder Condition | 12 weeks
Change from baseline to Week 4 and 12 in AUA Symptom Index | 12 weeks
Change from baseline to Week 4 and 12 in OAB questionnaire | 12 weeks
Clinical Global Impression-Improvement at Week 12 | 12 weeks
Overall Treatment Effect Scale of Overactive Bladder Control at Week 4 and 12 | 12 weeks
To asses the safety of tolterodine in patients with OAB | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (86):
- United States (86):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Sun Lakes, Arizona
  - Pfizer Investigational Site, Bentonville, Arkansas
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Buena Park, California
  - Pfizer Investigational Site, Foothill Ranch, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, West Covina, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Lakewood, Colorado
  - Pfizer Investigational Site, Chipley, Florida
  - Pfizer Investigational Site, Davie, Florida
  - Pfizer Investigational Site, Hallandale, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Miami Beach, Florida
  - Pfizer Investigational Site, Murdock, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Saint Cloud, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Barnesville, Georgia
  - Pfizer Investigational Site, Blue Ridge, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Naperville, Illinois
  - Pfizer Investigational Site, Orland Park, Illinois
  - Pfizer Investigational Site, Newton, Kansas
  - Pfizer Investigational Site, Shawnee Mission, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Marrero, Louisiana
  - Pfizer Investigational Site, Laurel, Maryland
  - Pfizer Investigational Site, Oxon Hill, Maryland
  - Pfizer Investigational Site, Jackson, Michigan
  - Pfizer Investigational Site, Portage, Michigan
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Blackwood, New Jersey
  - Pfizer Investigational Site, Mount Laurel, New Jersey
  - Pfizer Investigational Site, Binghamton, New York
  - Pfizer Investigational Site, Endicott, New York
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, Kingston, New York
  - Pfizer Investigational Site, Beaufort, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Morehead City, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Central Point, Oregon
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Bala-Cynwyd, Pennsylvania
  - Pfizer Investigational Site, Bensalem, Pennsylvania
  - Pfizer Investigational Site, Connellsville, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, Stoneboro, Pennsylvania
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Simpsonville, South Carolina
  - Pfizer Investigational Site, Cordova, Tennessee
  - Pfizer Investigational Site, Huntingdon, Tennessee
  - Pfizer Investigational Site, Lexington, Tennessee
  - Pfizer Investigational Site, Savannah, Tennessee
  - Pfizer Investigational Site, Selmer, Tennessee
  - Pfizer Investigational Site, Waynesboro, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Colleyville, Texas
  - Pfizer Investigational Site, Friendswood, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, West Jordan, Utah
  - Pfizer Investigational Site, West Valley City, Utah
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
  - Pfizer Investigational Site, New Berlin, Wisconsin
  - Pfizer Investigational Site, Oregon, Wisconsin
  - Pfizer Investigational Site, Wauwatosa, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121001&StudyName=A%20Study%20to%20Evaluate%20the%20Efficacy%20of%20Tolterodine%20on%20Specific%20Symptoms%20in%20Adult%20Patients%20with%20Overactive%20Bladder.%20